CLINICAL TRIAL: NCT01691001
Title: Effect of Dexmedetomidine on Sevoflurane Requirements and Emergence Agitation in Children Undergoing Ambulatory Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4-2011-0430
Record Dates: First submitted 2012-09-12; First posted 2012-09-24 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Ambulation Difficulty
MeSH Terms: conditions — Mobility Limitation | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- dexmedetomidine (Experimental)
  Interventions: Drug: Dexmedetomidine
- placebo group (Placebo Comparator): normal saline
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Dexmedetomidine — dexmedetomidine(vs saline) 1 mcg/kg iv bolus during 10minutes, and then, 0.1 mcg/kg/h dexmedetomidine(vs saline) was infused.
  Arms: dexmedetomidine
Drug: normal saline
  Arms: placebo group

SUMMARY:
Although the aetiology of emergence agitation (EA) derives from multiple factors, it is a frequent side effect of sevoflurane anaesthesia in children. Dexmedetomidine, a potent selective α2-adrenergic agonist, can reduce the doses of hypnotics, opioids, analgesics, and anaesthetics that must be concomitantly administered. This study was conducted to assess the effect of dexmedetomidine infusion on sevoflurane requirements and recovery profiles with EA in children undergoing ambulatory surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA class I
* obtaining written informed consent from the parents
* aged 1-5 years, and weighing <20 kg who were undergoing ambulatory hernioplasty or orchiopexy

Exclusion Criteria:

* mental retardation
* developmental delays
* neurological or psychiatric illnesses
* coagulation disorder
* spinal anomalies
* bilateral procedures

Ages: 1 Year to 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2011-08; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
the reduction rate of ET-sevo in achieving BIS scores from 45-50 | 2 hour(during whole operation period)

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seoul, South Korea